CLINICAL TRIAL: NCT05303623
Title: Radiological and Cardiopulmonary Evaluation of the Effect of Inspiratory Muscle Training on Diaphragmatic Function in Mechanically Ventilated Patients in the Intensive Care Unit
Brief Title: The Effect of Inspiratory Muscle Training on Diaphragmatic Function in Mechanically Ventilated Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Demiroglu Bilim University (Other)
Responsible Party: Principal Investigator, Reyhan Kaygusuz, Lecturer, Istanbul Demiroglu Bilim University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: doctoral thesis
Record Dates: First submitted 2022-03-22; First posted 2022-03-31 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Intensive Care Unit Acquired Weakness
Keywords: mechanical ventilated patients; Inspiratory muscle training; Physiotherapy and rehabilitation; diaphragmatic issue doppler; Respiratory muscle thickness

STUDY DESIGN:
Intervention Model Description: Parallel Assignment Randomized Healthy participants
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional Physiotherapy (Experimental): In the intensive care unit and who had mechanical ventilation for more than 48 hours and who were extubated. Medical, physical and respiratory examination in this group Physical Function Test in Intensive Care (PFIT), maximum inspiratory mouth pressure and maximum expiratory mouth pressure, Medical Research Council Muscle Strength Test and diaphragmatic function with B mode and M mode ultrasonographic assessment.
  In this group will apply only conventional physiotherapy. Conventional physiotherapy to contain breathing and,thoracal expansion exercises, bronchial hygiene techniques and gradual mobilization. Conventional physiotherapy apply for 5 days after extubation period 1 time a day.
  Interventions: Other: Conventional Physiotherapy
- Conventional Physiotherapy + inspiratory muscle training (Experimental): Physical ,medical and respiratory examination in this group Physical Function Test in Intensive Care (PFIT), maximum inspiratory mouth pressure and maximum expiratory mouth pressure, Medical Research Council Muscle Strength Test and diaphragmatic function with B mode and M mode ultrasonographic assessment. In this group, inspiratory muscle training will be applied in addition to conventional physiotherapy.
  Inspiratory muscle training apply for 5 days after extubation period. Inspiratory muscle training will be given with a threshold loading by giving resistance at 30-40% of the maximum inspiratory pressure measurement obtained. The subjects in this group will be given inspiratory muscle training 4 sets with 6-10 breaths per set, 1-2 minutes between each set once a day in addition to conventional physiotherapy.
  Interventions: Other: Conventional Physiotherapy+ inspiratory muscle training
- Healthy Subject (Experimental): In the group consisting of healthy volunteers, which will be taken to determine the normative values of the outcome measurements for diaphragmatic tissue Doppler imaging and ultrasonographic evaluation, 2 sessions a day with a threshold-loaded inspiratory muscle training device, starting at 30% of the MIP value, 5 days a week for 4 weeks. Inspiratory muscle training will be performed in 4 sets, 6-8 breaths in each set and 2 minutes rest between sets. In the second evaluation to be made after the inspiratory muscle training, the above-mentioned evaluations and measurements will be repeated.
  Interventions: Other: inspiratory muscle training

INTERVENTIONS:
Other: Conventional Physiotherapy — Conventional Physiotherapy to contain breathing and thoracal expansion exercises, bronchial hygiene techniques and gradual mobilization in 1 time a day.
  Arms: Conventional Physiotherapy
Other: Conventional Physiotherapy+ inspiratory muscle training — Conventional Physiotherapy to contain breathing and thoracal expansion exercises, bronchial hygiene techniques and gradual mobilization in 1 time a day. In this group addition to conventional physiotherapy inspiratory muscle training will be performed with the threshold-loaded inspiratory muscle training device, starting at 30% of the maximum inspiratory mouth pressure value, during 5 days, in 2 sessions, 4 sets per day, 6-8 breaths in each set and 2 minutes of rest between sets.
  Arms: Conventional Physiotherapy + inspiratory muscle training
Other: inspiratory muscle training — In this group inspiratory muscle training will be performed with the threshold-loaded inspiratory muscle training device, starting at 30% of the maximum inspiratory mouth pressure value, during 5 days, in 2 sessions, 4 sets per day, 6-8 breaths in each set and 2 minutes of rest between sets.
  Arms: Healthy Subject

SUMMARY:
In this study, the effect of inspiratory muscle training on diaphragmatic functions will be investigated radiologically in mechanically ventilated patients.

DETAILED DESCRIPTION:
Many patients who receive treatment in intensive care need mechanical ventilation support. Invasive mechanical ventilation is an application used in critically ill patients to provide pulmonary gas exchange and to relieve the respiratory muscles. Mechanical ventilation and long- term bed rest induced extremity muscle weakness is a common condition in patients hospitalized in the intensive care unit. Acquired muscle weakness in intensive care is associated with poor prognosis and high mortality At the same time, mechanical ventilation can lead to the development of respiratory muscle dystrophy and atrophy.

Recently, a similar concern has arisen about the potential negative effects of mechanical ventilation on respiratory muscles. This condition is called ventilator-induced diaphragmatic dysfunction In patients with mechanical ventilation, dysfunction, muscle fiber type change and barotrauma are seen especially in the diaphragm, which is the primary inspiratory muscle. Diaphragmatic dysfunction may promote prolong of intubation, weaning difficulties and risk of increase reintubation in patients who are mechanically ventilated.

The effect of inspiratory muscle training, which is applied in addition to conventional respiratory physiotherapy, on diaphragmatic dysfunction, on the weaning process and the long of stay in intensive care has not been fully elucidated, and a limited number of studies have been conducted on this subject It has been reported that in patients with prolonged mechanical ventilation, diaphragmatic peak contraction velocity, peak relaxation velocity, movement speed, velocity time integral are lower than healthy individuals and this is correlated with failure to wean from mechanical ventilation. We could not find any report and clinical trial in the literature evaluation the effect of conventional physiotherapy and additional inspiratory muscle training on diaphragmatic tissue movement velocity and diaphragm thickness using detailed radiological methods in intensive care patients dependent on mechanical ventilation. In this context, our not working has a unique value. Our study will contribute to elucidating the mechanisms that affect the weaning process from mechanical ventilation in intensive care patients. It is aimed to develop strategies that will shorten the long of stay in intensive care and total hospital stay with therapeutic approaches that enable patients to be extubated as early as possible.

ELIGIBILITY:
For Patients Group Inclusion Criteria:

* Needing mechanical ventilation support longer than 2 days,
* Alert and Riker Sedation Agitation Score >4
* Being hemodynamically stable (HR<140 beats/min, BP stable)
* Dobutamine and minimal vasopressor use
* Fever of 36.5-38.5
* Body Mass Index <40 m2/cm,
* FiO2 of 0.5 or less,
* Absence of myocardial ischemia.

For Patients Group Exclusion Criteria:

* Noncooperation
* Phrenic nerve damage
* Chest wall trauma and/or deformity to prevent diaphragmatic movement
* Progressive neuromuscular disease with respiratory involvement
* There is enough secretion to require more than one aspiration every hour.
* Patients using sedative drugs continuously
* High-dose cortisol use
* Using a home mechanical ventilator before mechanical ventilation in intensive care unit

For Healthy Group Inclusion Criteria:

* With the control and intervention group, age, characteristics and characteristics,
* Chronic system and no ongoing treatment,
* Body mass index not 40 kg/m2,
* 18-80 years old

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-12-25 (Actual)

PRIMARY OUTCOMES:
Maximal inspiratory and expiratory pressure | Change from baseline Maximal inspiratory and expiratory pressure at 5th day
  Intraoral pressures measured at maximal respiration against a valve that closes the airway during maximal inspiration pressure and expiration. Maximal inspiration pressure is the highest pressure created to open closed alveoli at the residual volume level. In our study, respiratory muscle strength will be performed using a portable, electronic mouth pressure measuring with device. For the test, the applied person is given maximum expiration and at the end of this, the airway is closed with a valve and the person is asked to make maximum inspiration and continue it for 1-3 seconds. In the maximal expiration pressure measurement, after maximal inspiration, the person is asked to make a maximal expiration for 1-3 seconds against the closed airway. The best of the three measurements is selected. There should be no more than 10% or more than 10 cmH2O difference between the two best measured
Diaphragmatic B mode, M mode and Tissue Doppler Ultrasonographic Imagining | Change from baseline diaphragmatic evaluation at 5th day
  Doppler Ultrasound evaluation to evaluate the diaphragmatic tissue waveform will be performed with an ultrasound probe placed in the right hemidiaphragm. Tissue movement rates will be evaluated during inspiration and expiration. The maximum contraction and relaxation rate of the diaphragm will be recorded with the sonographic evaluation to be made during 10 normal breaths. In addition, while sitting upright with a 90 degree angle in two-dimensional B mode, diaphragm thickness will be measured from the right intercostal area from the midaxillary level, from the right subcostal area from the anterior axillary level and mid-clavicular level with the superficial probe during deep inspiration and deep expiration. Diaphragm mobility in normal inspiration and deep inspiration from the mid-axillary level from the right subcostal area with M-mode ultrasonography will be evaluated by a pulmonologist before and after the training.
Respiratory Muscle Thickness | Change from baseline Respiratory Muscle Ultrasonographic Imagining evaluation at 5th day
  With B mode ultrasound, the thickness of the internal oblique abdominis, external oblique abdominis and transversus abdominis muscles is measured 2-3 fingers above the umbilicus.
Physical Function Test (PFIT) battery | Change from baseline Physical Function Test (PFIT) battery 5th day
  The physical function levels of the cases in the intensive care unit will be evaluated with the Physical Function Test (PFIT) battery in the intensive care unit. PFIT is a test battery applied by the researcher, consisting of 4 main headings: Support (Stand up without sitting)', 'Cadence (steps/minute)', 'Shoulder (flexion strength)' and 'Knee (extension strength)'. are scored according to the degree of assistance (0-unassisted, 1-with the help of one person, 2-with the help of two people). Standing will be recorded as the number of steps and time performed in standing-stand action. Shoulder and knee muscle strength manual muscle test (0-unable , 1- there is only contraction, 2- completes the movement when gravity is eliminated, 3- completes the movement against gravity, 4- completes the movement with less than maximum resistance to gravity, 5- completes the movement with maximum resistance against gravity).
Medical Research Council(MRC) Strength Test | Change from baseline Medical Research Council(MRC) Strength Test battery 5th day
  Six muscle groups (abduction of the arm, flexion of the forearm, extension of the wrist, flexion of the hip, extension of the knee, and dorsal flexion of the foot) bilaterally. The tests were performed in the ICU. All muscle groups were scored between 0 and 5 (0 = no visible/palpable contraction; 1 = visible/palpable contraction without movement of the limb; 2 = movement of the limb but not against gravity; 3 = movement against gravity (almost full passive range of motion) but not against resistance; 4 = movement against gravity and resistance, arbitrarily judged to be submaximal for gender and age; 5 = normal).
Acute Care Index of Function (ACIF) | Change from baseline Acute Care Index of Function (ACIF) 5th day
  Sub-components of the ACIF include 'Mental Status,' 'Bed Mobility,' 'Transfers' and 'Mobility.'20 total item instrument with activities to measure cognition and functional mobility.

CONTACTS AND LOCATIONS:
Overall Officials: Barış Yılmaz, Specialist, Study Chair — Sureyyapasa Chest Diseases and Thoracic Surgery Training and Research Hospital
Locations (1):
- Istanbul Demiroglu University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No